CLINICAL TRIAL: NCT05175066
Title: Can Bisoprolol Administration Prevent Anthracycline-induced Cardiotoxicity?: a Double-blind Randomized Trial.
Brief Title: Bisoprolol Administration to Prevent Anthracycline-induced Cardiotoxicity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Manoochehr Ebrahimian, Principal Investigator, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SamanRostambeigi
Record Dates: First submitted 2021-12-24; First posted 2022-01-03 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Cardiomyopathies; Chemotherapy Effect; Diastolic Dysfunction; Systolic Dysfunction
Keywords: Bisoprolol; Cardiomyopathy; Chemotherapy; Anthracyclines
MeSH Terms: conditions — Cardiomyopathies | interventions — Bisoprolol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bisoprolol (Experimental): 40 patients who were given bisoprolol at a dose of 1.25 mg daily, and in the absence of clinical symptoms and heart rate above 60 and systolic blood pressure above 100, 1.25 mg was added to the therapeutic dose every 2 weeks to reach 5 mg daily.
  Interventions: Drug: Bisoprolol
- Placebo (Placebo Comparator): Two placebo tablets in similar shape and color to bisoprolol were given on a daily basis to each of the 40patients as the control group.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bisoprolol — For patients who were candidates to start therapy with anthracycline, bisoprolol was administrated as explained before to determine the effect of this drug on the reduction of anthracycline-induced cardiomyopathy.
  Arms: Bisoprolol
Drug: Placebo — Tablets with similar shape and size and color to bisoprolol were given to the patients whom undergone chemotherapy with anthracyclines to compare the effects between two groups.
  Arms: Placebo

SUMMARY:
Anthracyclines are one of the most well-known and effective drugs used to treat malignancies.The most important limiting factor in the use of this drug is its cardiac toxicity which includes cardiomyopathy and congestive heart failure. Bisoprlol is a β1-specific β-blocker that can reduce cardiac overload and also have anti-inflammatory antioxidant effects and can reduce reactive oxygen metabolites so it can be used as a cardioprotective agent in patients with a high risk of heart failure. To the best of our knowledge, no study has been performed to evaluate the prophylactic effect of bisoprolol solely in patients under chemotherapy with anthracyclines. This study is aimed to evaluate the cardioprotective role of bisoprolol in patients with non-metastatic breast cancer receiving doxorubicin, by measuring global longitudinal strain before and after treatment.

DETAILED DESCRIPTION:
This study was a double-blinded randomized control trial that was conducted at the Iran University of medical sciences.

Sixty-three patients that was diagnosed with non-metastatic breast cancer and anthracycline-based chemotherapy were planned for them were enrolled in this study. The exclusion criteria included: established ischemic heart disease, baseline LVEF <50%, cardiomyopathy (restrictive, dilated, or hypertrophic) detected by transthoracic echocardiography, moderate or severe valvular disease, prior chemotherapy, presence of contraindication for beta-blockers and cardiac arrhythmias and lack of patient compliance. Also, all the patients that had consumed angiotensin-converting enzyme Inhibitors, angiotensin receptor Inhibitors,diuretics, statins,other beta-blockers or non-dihydropyridin calcium channel blockers were excluded.Pateinets were randomly divided into two case and control groups by a box randomization method. At first, case group was comprised of 31 patients who were given bisoprolol at a dose of 1.25 mg daily, and in the absence of clinical symptoms and heart rate above 60 and systolic blood pressure above 100, 1.25 mg was added to the therapeutic dose every 2 weeks to reach 5 mg daily.

Two placebo tablets in similar shape and color to bisoprolol were given on a daily basis to each of the remaining 32 patients as the control group. Both bisoprolol and placebo administration was started since 7 days before start of chemotherapy and continued for 6 months.The study protocol was explained to each patient, and written consent was obtained from all patients.

chemotherapy regimen included doxorubicin (60 mg/m 2) and cyclophosphamide (600 mg/m2) followed by docetaxel (100 mg/m2) that was completed in four consecutive cycles, each cycle lasted 21 days and the cumulative dose of doxorubicin reached 240 mg/m2.

None of patients were treated with hormonal therapy or trastuzumab during the study period. Patients were visited by a cardiologist at baseline, before chemotherapy and every month after start of treatment. The presence of drug-related side effects (in particular hypotension and bradycardia) if any were recorded. The occurrence of heart failure, hospitalization and death were also collected.

Transthoracic echocardiography was performed 1 week prior to the chemotherapy and 1 week after the fourth doxorubicin cycle. Strain, strain-rate parameters and LVEF wereevaluated. A decrease of more than 10-50% in LVEF was considered as a criterion for discontinuing chemotherapy with anthracycline and patients were excluded from the study.

Blind conventional 2D echocardiography done using an EPIQ 7 premium ultrasound system (Philips Healthcare, Stockholm, Sweden) equipped with a 2.5-MHz transducer. All measurements were performed following the recommendations of the American Society of Echocardiography (21)in apical (2- and 4-chamber and apical long axis) and parasternal (long and short axis) views and measured at the time of acquisition without reference to previous measurements. Images was digitally stored for off-line Speckle-tracking analysis (EchoPAC 108.1.5, GE-Vingmed). Longitudinal strain, evaluating the shortening (negative strain) and lengthening (positive strain) of the myocardial wall, was measured from the three apical views (long-axis and two- and four-chamber views): GLS was calculated by averaging the peak strain values of 18 segments. The mean frame rate of 2D images was 90 ±4 frames/s.

SPSS version 18.0 (SPSS, Inc., Chicago, IL) was used for statistical analysis. All quantitative data have been expressed as mean ± SD.Categorical variables were summarized as number(percent), and continuous variables as either median (range) or mean ± standard deviation. Independent-sample t-tests were used to compare LVEF, strain and strain-rate parameters between the two groups before and after the intervention. Paired sample t-tests were used to compare the echocardiography findings in each group before and after the chemotherapy. P-values less than 0.05 were considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

patients that was diagnosed with non-metastatic breast cancer and anthracycline-based chemotherapy were planned for them

Exclusion Criteria:

* Established ischemic heart disease
* Baseline LVEF <50%, cardiomyopathy (restrictive, dilated or hypertrophic) detected by transthoracic echocardiography
* Moderate or severe valvular disease,
* Prior chemotherapy,
* Presence of contraindication for beta-blockers and cardiac arrhythmias and lack of patient compliance
* Patients that had consuming angiotensin converting enzyme Inhibitors, angiotensin receptor Inhibitors,diuretics,statins,other beta-blockers or non-dihydropyridin calcium channel blockers

Ages: 35 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with Non-metastatic breast cancer that undergone Anthracyclin-based chemotherapy regimen
Enrollment: 80 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-10-07 (Actual); Study Completion 2021-12-02 (Actual)

PRIMARY OUTCOMES:
LVEF | Baseline and after 6 months
  Change in Left ventricular ejection-fraction after chemotherapy
GLS | Baseline and after 6 months
  Change in global longitudinal strain after chemotherapy

SECONDARY OUTCOMES:
Diastolic dysfunction | Baseline and after 6 months
  Occurrence of diastolic dysfunction after chemotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Rasool Akram hospital, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes
All the data and analytic works will be available for interested persons.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From February 2022
Access Criteria: Everyone with verified institutional email.

REFERENCES:
- [Background] Tashakori Beheshti A, Mostafavi Toroghi H, Hosseini G, Zarifian A, Homaei Shandiz F, Fazlinezhad A. Carvedilol Administration Can Prevent Doxorubicin-Induced Cardiotoxicity: A Double-Blind Randomized Trial. Cardiology. 2016;134(1):47-53. doi: 10.1159/000442722. Epub 2016 Feb 12. PMID 26866364
- [Background] Silber JH, Cnaan A, Clark BJ, Paridon SM, Chin AJ, Rychik J, Hogarty AN, Cohen MI, Barber G, Rutkowski M, Kimball TR, Delaat C, Steinherz LJ, Zhao H. Enalapril to prevent cardiac function decline in long-term survivors of pediatric cancer exposed to anthracyclines. J Clin Oncol. 2004 Mar 1;22(5):820-8. doi: 10.1200/JCO.2004.06.022. PMID 14990637